CLINICAL TRIAL: NCT06190366
Title: Effects of Bloodletting Acupuncture for Subacute and Chronic Non-specific Low Back Pain - a Randomized Controlled Trial
Brief Title: Effects of Bloodletting Acupuncture for Subacute and Chronic Non-specific Low Back Pain
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Charite University, Berlin, Germany (Other)
Responsible Party: Principal Investigator, Andreas Michalsen, Principal Investigator, Charite University, Berlin, Germany
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Mikroaderlass
Record Dates: First submitted 2023-12-19; First posted 2024-01-05 (Actual); Last update posted 2024-01-05 (Actual); Status verified 2024-01

CONDITIONS: Back Pain, Low
MeSH Terms: conditions — Low Back Pain

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Bloodletting acupuncture at the fossa poplitea (Experimental)
  Interventions: Procedure: Bloodletting acupuncture at the fossa poplitea
- Bloodletting acupuncture at the regio glutaea (Experimental)
  Interventions: Procedure: Bloodletting acupuncture at the regio glutaea
- Waiting list control group (No Intervention)

INTERVENTIONS:
Procedure: Bloodletting acupuncture at the fossa poplitea — This group is treated with bloodletting acupuncture at the fossa poplitea. The treatment takes place twice a week from week 1 to week 3. This means that 6 treatments of approx. 20 minutes each should be carried out within the 3 weeks.
  Arms: Bloodletting acupuncture at the fossa poplitea
Procedure: Bloodletting acupuncture at the regio glutaea — This group is treated with bloodletting acupuncture at the regio glutaea. The treatment takes place twice a week from week 1 to week 3. This means that 6 treatments of approx. 20 minutes each should be carried out within the 3 weeks.
  Arms: Bloodletting acupuncture at the regio glutaea

SUMMARY:
Evaluation of a bloodletting acupuncture at the fossa poplitea in comparison to bloodletting acupuncture at the regio glutaea and a waiting list control group in patients with subacute and chronic non-specific pain low back pain.

ELIGIBILITY:
Inclusion Criteria:

* Specialist confirmed diagnosis of subacute or chronic non-specific low back pain for at least 6 weeks prior to inclusion
* Average pain intensity with at least 50 mm on the VAS from 0 to 100 mm

Exclusion criteria:

* Serious illnesses
* Poor general condition
* Coagulation disorder, therapy with anticoagulants
* Thrombophlebitis, skin inflammation in the area of the lower extremities
* Alcohol, drug or medication addiction
* Pregnancy
* Lack of willingness to cooperate, linguistically or mentally unable to understand the contents of the study
* Participation in another clinical trial during the study period
* Starting a new therapy for the treatment of low back pain in the last 2 weeks

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 108 (Estimated)
Dates: Start 2023-12-19 (Actual); Primary Completion 2024-12 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Change from baseline in average pain intensity in previous week | Baseline, 3 weeks
  Intensity of pain in previous week as measured on a 100 mm visual analog scale (0-100).

SECONDARY OUTCOMES:
Change from baseline in average pain intensity in previous week | Baseline, 6 weeks
  Intensity of pain in previous week as measured on a 100 mm visual analog scale (0-100).
Change from baseline in average pain intensity of the last 24 hours | Baseline, 3 weeks, 6 weeks
  Intensity of pain in previous week as measured on a 100 mm visual analog scale (0-100).
Change from baseline for back pain specific disability | Baseline, 3 weeks, 6 weeks
  Use of standardized Roland Morris Disability Questionnaire (RMDQ) to assess back pain specific disability. The scale ranges from 0 to 100, where 0 is the lowest level and 100 is the highest level.
Change from baseline in pain bothersomeness in previous week | Baseline, 3 weeks, 6 weeks
  Bothersomeness in previous week as measured on a 100 mm visual analog scale (0-100).
Change from baseline for days with pain medication use | Baseline, 3 weeks, 6 weeks
  Specific self-reported pain medication use
Change from baseline for health related quality of life | Baseline, 3 weeks, 6 weeks
  Use of standardized Short Form 36 Health Survey (SF-36). The scale ranges from 0 to 100, where 0 is the lowest level and 100 is the highest level.
Change from baseline for pain self-efficacy | Baseline, 3 weeks, 6 weeks
  Use of standardized Pain Self-Efficacy Questionnaire (PSEQ). The scale ranges from 0 to 100, where 0 is the lowest level and 100 is the highest level.
Change from baseline for anxiety and depression | Baseline, 3 weeks, 6 weeks
  Use of standardized Hospital Anxiety and Depression Scale (HADS). The scale ranges from 0 to 100, where 0 is the lowest level and 100 is the highest level.
Change from baseline for work productivity | Baseline, 3 weeks, 6 weeks
  Use standardized Work Productivity and Activity Impairment Questionnaire (WPAI) to assess employment status and productivity. The scale ranges from 0 to 100, where 0 is the lowest level and 100 is the highest level.

OTHER OUTCOMES:
Number of participants with adverse events as a measure of safety and treatment adherence | 3 weeks, 6 weeks
  Identify and assess self reported and unanticipated adverse events over the course of the study as a measure of safety and treatment adherence.
Treatment adherence | 3 weeks
  Assess treatment adherence according to attendance during 3 week intervention period.
Treatment expectation: effectiveness of bloodletting acupuncture in reducing low back pain | Baseline
  Assess treatment expectation at baseline, Likert scale (1-very good effectiveness to 5-poor effectiveness)

CONTACTS AND LOCATIONS:
Locations (1):
- Charité Hochschulambulanz für Naturheilkunde, Immanuel Krankenhaus Berlin, Berlin, Germany

IPD SHARING:
Plan to Share IPD: No